CLINICAL TRIAL: NCT05900037
Title: A Prospective, Multicenter, Randomized Clinical Investigation Evaluating GATT-Patch for Hemostasis During Minimally Invasive Liver and Gallbladder Surgery
Brief Title: GATT-Patch Versus SURGICEL® Original in Minimally Invasive Liver and Gallbladder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GATT Technologies BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DHF-01-SP-065
Record Dates: First submitted 2023-05-19; First posted 2023-06-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Intraoperative Bleeding; Liver Diseases; Gallbladder Diseases; Hemorrhage, Surgical
Keywords: Hemostatic patch; GATT-Patch; SURGICEL® Original; Liver surgery; Gallbladder surgery; Hemostasis
MeSH Terms: conditions — Blood Loss, Surgical; Liver Diseases; Gallbladder Diseases

STUDY DESIGN:
Intervention Model Description: Randomization 1:1
Who Masked: Participant
Masking Description: Patients will be blinded to randomized treatment and treatment used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- GATT-Patch (Experimental): Hemostatic Patch
  Interventions: Device: GATT-Patch
- SURGICEL® Original (Active Comparator): Hemostatic Patch
  Interventions: Device: SURGICEL® Original

INTERVENTIONS:
Device: GATT-Patch — GATT-Patch is a sterile, flexible and resorbable hemostatic sealing patch. It presents as a blue, soft, flexible, porcine gelatin fiber-based carrier impregnated with an NHS-POx / NU-POx granulate. GATT-Patch measures 10 cm long by 5 cm wide. GATT-Patch is active and can be applied on both sides. Blue color is an aid to visualize GATT-Patch when applied onto a bleeding location.
  GATT-Patch is indicated for use as an adjunct to hemostasis in surgery for minimal, mild or moderate bleeding sites when control of bleeding by standard surgical techniques (such as suture, ligature or cautery) is ineffective or impractical. GATT-Patch is intended to be used for management of hemorrhage during surgeries on the liver.
  Arms: GATT-Patch
Device: SURGICEL® Original — SURGICEL® Absorbable Hemostat (oxidized regenerated cellulose) is indicated for use in surgical procedures to assist in the control of capillary, venous and small arterial hemorrhage when ligation or other conventional methods of control are impractical or ineffective.
  Other Names: Surgicel Absorbable Hemostat
  Arms: SURGICEL® Original

SUMMARY:
This is a pre-market, prospective, randomized (1:1), multicenter, pivotal clinical investigation. The purpose of this investigation is to determine the clinical performance of GATT-Patch as compared with SURGICEL® Original for the management of minimal, mild, or moderate bleeding during minimally invasive liver and gallbladder surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled to undergo elective minimally invasive (robotic or laparoscopic) surgery on the liver, including cholecystectomy
* Subject is willing and able to give written informed consent for the clinical investigation participation
* Subjects is 22 years of age or older at the time of enrollment; and
* Subject has been informed of the nature of the clinical investigation.

A subject must meet all of the following intra-operative inclusion criteria to be enrolled into the clinical investigation:

* Subject undergoes a fully minimally invasive surgical approach without the use of a hand port at the time of randomization and application of the patch;
* Subject in whom the Investigator is able to identify a target bleeding site at the liver resection plane for which any applicable conventional means for hemostasis (e.g. suture, ligature or cautery) are ineffective or impractical, and the choice is made to use a hemostatic agent to stop the bleeding
* Pressure on the surface of the hemostatic agent can be applied with the minimally invasive instruments to achieve hemostasis
* Subject has a target bleeding site with a SBSS of 1, 2, or 3 (e.g. reflecting minimal, mild or moderate bleeding severities)

Exclusion Criteria:

* The target bleeding site is from a large defect in an artery or vein that requires vascular reconstruction with maintenance of vessel patency
* Subject is scheduled to undergo surgery on organs other than the liver and its associated biliary and vascular system
* Subject is scheduled to undergo a staged liver surgery procedure (e.g., Associating Liver Partition and Portal vein ligation for Staged hepatectomy [ALPPS])
* Subject is taking multiple antithrombotic therapies in therapeutic dosage up to the time of surgery, but allowing exclusive use of acetylsalicylic acid
* Subject has platelet count <100 x 109/L, an activated partial thrombin time of >100s, or international normalized ratio >2.5
* Subject has a total bilirubin level of ≥2.5 mg/dl
* Subject is pregnant, planning on becoming pregnant or actively breastfeeding during the 3-month follow-up period
* Subject has a known hypersensitivity to brilliant blue (FD&C Blue #1), porcine gelatin
* Subject who has religious objections to receiving products containing porcine
* Subject has an active or suspected infection at the bleeding site
* Subject in whom the investigational device will be used at the site of a synthetic graft or patch implant
* Subject has a life expectancy of less than 3 months
* Subject has a documented severe congenital or acquired immunodeficiency
* Subject has had or has planned to receive any organ transplantation
* Subject undergoes surgery with the indication of being a living liver donor
* Subject is currently participating or has participated in another clinical investigation within the past 30 days that may affect the endpoints of the study, such as trials related to the surgical procedure and anti-coagulation
* Subject is not appropriate for inclusion in the clinical investigation, per the medical opinion of the Investigator
* Subject has any incidental (pre- and peri-operative) findings deemed by the Investigator to potentially jeopardize the safety or welfare of the subject

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Rate of hemostasis within 7 minutes from introduction of the first (piece of) patch through the trocar without rebleeding at the 10-minute time point from initiating pressure on the entire surface of the hemostatic agent | During surgical procedure
  SBSS 0

SECONDARY OUTCOMES:
Median time in seconds from introducing the hemostatic agent through the trocar and achieving hemostasis | During surgical procedure
  SBSS 0
Median time in seconds from introducing the hemostatic agent through the trocar to initiating pressure on the entire surface of the agent | During surgical procedure
  SBSS 0
Median time in seconds to hemostasis from initiating pressure on the entire surface of the agent | During surgical procedure
  SBSS 0
Percentage of hemostasis from initiating pressure on the entire surface of the agent at 30, 60, 120, 180, 240, 300, 360, 420, 480, 540 and 600 seconds | During surgical procedure
  SBSS 0-5
Kaplan-Meier estimated distribution of time to hemostasis from initiating pressure on the entire surface of the agent | During surgical procedure
  SBSS 0
Treatment failure, defined as no hemostasis with the agent at 10 minutes from initiating pressure on the entire surface of the agent | During surgical procedure
  SBSS 1-5 at the 10 minute timepoint
Rebleeding after the 10-minute time point from initiating pressure on the entire surface of the agent but before subject wound closure | During surgical procedure
  SBSS 1-5 after initially SBSS 0
Number of times an additional (piece of) hemostatic agent needs to be used to achieve hemostasis | During surgical procedure
  SBSS 1-5

OTHER OUTCOMES:
Conversion from minimally invasive to open surgery, and reasons for conversion | During surgical procedure
  SBSS 1-5
Procedure duration | During surgical procedure
  Time in minutes
Duration of hepatic blood inflow reduction | During surgical procedure
  Time in minutes
Estimated blood loss during surgery | During surgical procedure
  mL
Number and type of blood transfusions during hospitalization | During surgical procedure
  Platelets, Erythrocytes, Plasma
Duration of Intensive Care Unit (ICU) stay | During hospitalization up to hospital discharge after the surgical procedure, estimated up to 30 days
  Time in Days
Total hospitalization time | From surgery to discharge from the ICU, estimated up to 30 days
  Time in Hours
Postoperative drainage volume, characteristics, and duration | During hospitalization up to hospital discharge after the surgical procedure, estimated up to 30 days
  Serous, sanguineous, serosanguineous, other Sanguineous Serosanguinous Serous, Sanguineous, Serosanguineous, Purulent, Other
Rate of subjects requiring reoperation | During postoperative 3-months follow-up
  Occurrence yes/no
Rate of subjects with liver resection surface complications on ultrasound | At 6 week follow-up visit
  Fluid collection, biloma, hematoma, patch encapsulation, patch rolling up on the surface
Amount of hemostatic material needed versus bleeding surface | During surgical procedure
  cm2 patch per cm2 bleeding
GATT-Patch device-specific user satisfaction questionnaire | At completion of the surgical procedure, at day 0
  Likert scale (strongly disagree, disagree, neutral, agree, strongly agree) with (strongly) agreeing meaning a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Head, MD PhD, Study Director — GATT Technologies BV
Locations (6):
- United States (6):
  - University of Southern California, Los Angeles, California
  - Washington University, St Louis, Missouri
  - Capital Health, Pennington, New Jersey
  - Weill-Cornell, New York, New York
  - Atrium Health, Charlotte, North Carolina
  - Intermountain Healthcare, Murray, Utah

IPD SHARING:
Plan to Share IPD: Yes
Undecided

REFERENCES:
- [Background] Boerman MA, Roozen E, Sanchez-Fernandez MJ, Keereweer AR, Felix Lanao RP, Bender JCME, Hoogenboom R, Leeuwenburgh SC, Jansen JA, Van Goor H, Van Hest JCM. Next Generation Hemostatic Materials Based on NHS-Ester Functionalized Poly(2-oxazoline)s. Biomacromolecules. 2017 Aug 14;18(8):2529-2538. doi: 10.1021/acs.biomac.7b00683. Epub 2017 Jul 25. PMID 28699748
- [Background] Roozen EA, Warle MC, Lomme RMLM, Felix Lanao RP, van Goor H. New polyoxazoline loaded patches for hemostasis in experimental liver resection. J Biomed Mater Res B Appl Biomater. 2022 Mar;110(3):597-605. doi: 10.1002/jbm.b.34938. Epub 2021 Sep 18. PMID 34536065